CLINICAL TRIAL: NCT03309449
Title: A Usability Assessment of Intramuscular, Atomized Intranasal, and Nasal Spray Administration of Naloxone by Community Members
Brief Title: A Usability Assessment of Naloxone by Community Members
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 922070-1
Record Dates: First submitted 2016-07-11; First posted 2017-10-13 (Actual); Results first posted 2021-11-02 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Drug Overdose
MeSH Terms: conditions — Drug Overdose | interventions — Syringes; Needles; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Intramuscular administration (Other): Participants in this arm will be provided with the training and supplies to administer intramuscular simulated naloxone using a syringe and needle to a simulated flesh pad on a mannequin.
  Interventions: Device: Syringe and needle
- Intranasal (Atomizer) (Other): Participants in this arm will be provided with the training and supplies to administer atomized intranasal simulated naloxone to a mannequin via a syringe using an intranasal mucosal atomization device.
  Interventions: Device: Intranasal mucosal atomization device
- Intranasal (Spray) (Other): Participants in this arm will be provided with the training and supplies to administer an intranasal spray simulated naloxone to a mannequin.
  Interventions: Device: Nasal spray

INTERVENTIONS:
Device: Syringe and needle — Intramuscular administration of simulated naloxone
  Arms: Intramuscular administration
Device: Intranasal mucosal atomization device — Intranasal atomizer administration of simulated naloxone
  Arms: Intranasal (Atomizer)
Device: Nasal spray — Nasal spray administration of simulated naloxone
  Arms: Intranasal (Spray)

SUMMARY:
This will be a usability trial to assess administration of naloxone via intramuscular, atomized intranasal, and nasal spray routes by nonmedical community members. Participants will undergo blocked randomization to naloxone kits containing supplies for one of the aforementioned routes and view an instructional video on how to appropriately administer the kit they were assigned. Participants will then have the opportunity to administer the simulated drug to a mannequin designated to simulate the route of administration assigned to the participant. The rate of successful administration will be determined for each route.

DETAILED DESCRIPTION:
Objectives:

* Primary: The successful administration of simulated naloxone. A successful administration will be defined as administration of the simulated naloxone to the mannequin head or simulated flesh pad within 10 minutes and without any critical errors (defined below).
* Secondary: Total time required to successfully administer the simulated naloxone.

Design: Single site, open-label, randomized usability assessment of intramuscular, intranasal, and nasal spray administration of simulated naloxone. A convenience sample of participants will consent to volunteer in the study at a public venue. Participants will provide verbal consent and will be randomly assigned a simulated naloxone kit containing either intramuscular, intranasal, or nasal spray administration materials. Participants will be shown an instructional video demonstrating how to appropriately assemble and administer the simulated naloxone kit they were randomly assigned. Once the video is complete the individual will enter a use scenario station where they will be asked to assemble and administer the simulated naloxone kit to a mannequin (intranasal and nasal spray) or simulated flesh pad (intramuscular). The participant will be instructed to start and will be timed until the simulated naloxone has been successfully administered or 10 minutes has elapsed. The participant will be observed by one trained investigator who will assess for successful administration of the simulated naloxone and critical errors. The environment will contain distractors (radio playing) and items that will simulate a community based dwelling (table, chairs, and an inflatable mattress). The mannequin and simulated flesh pad will be located on the mattress. Once the participant has successfully administered simulated naloxone or 10 minutes elapses the timer will be stopped. Successful administration of simulated naloxone will be defined as administration of the agent without any critical errors occurring (defined below). Data collected will include demographics (defined below), successful administration of simulated naloxone, and time to successful administration of simulated naloxone.

Statistical Methods: All data will be analyzed using IBM SPSS Statistics software. Demographics data will be analyzed using descriptive statistics for continuous measures and percentages for categorical measures. The successful administration of naloxone will be compared between groups using the Chi-square test and a significant difference will be defined as a p-value of less than 0.05 for the result. The time to administration between groups will be assessed using a one-way ANOVA and a significant difference will be defined as a p-value of less than 0.05 for the result.

Data Analysis/Interpretation: As stated above data will be collected to assess both the successful administration of and time to administration of naloxone. The rate of successful administration will be reported as a percentage for each of the three groups and analyzed using the Chi-square test. Successful administration is defined as administration of the simulated naloxone within 10 minutes without committing any critical errors. Critical errors are as follows:

* Intranasal (atomizer): failure to remove both yellow caps from bristoject, failure to remove cap from simulated naloxone, failure to attach atomizer, failure to attach simulated naloxone, drug leak prior to administration, administration in only one nostril, and failure to administer within 10 minutes.
* Intramuscular: failure to attach the needle to the syringe, failure to remove cap from simulated naloxone, failure to draw up >90% (0.9 mL) of the simulated naloxone, failure to puncture simulated flesh pad with needle, failure to push entire volume of fluid in the syringe into the simulated flesh pad, and failure to administer within 10 minutes.
* Intranasal (spray): failure to place the tip of the device into one nostril, failure to depress the device and release the simulated naloxone, failure to administer within 10 minutes.

Time to successful administration will be reported using descriptive statistics (mean time to administration) and analyzed using a one-way ANOVA. Times for participants who commit a critical error or who do no administer the simulated naloxone within 10 minutes will not be included in the analysis.

A route of administration will be considered to be more user-friendly if it demonstrates a statistically significantly higher rate of successful administration compared to another route of administration.

Study Procedures: No study procedures will be performed on study participants.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults at least 18 years of age

Exclusion Criteria:

* severely visually or hearing impaired (defined as: legally deaf, legally blind, unable to read print size provided on instructional handout, or unable to hear video audio), previous naloxone administration training, not English proficient, previously participated in the trial, or pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Eggleston, PharmD, Principal Investigator — State University of New York - Upstate Medical University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intramuscular Administration | Intranasal (Atomizer) | Intranasal (Spray)
Started | 46 | 46 | 46
Completed | 46 | 46 | 46
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intramuscular Administration | Intranasal (Atomizer) | Intranasal (Spray) | Total
Number analyzed (Participants) | 46 | 46 | 46 | 138
Age, Continuous [Median (Full Range); unit: Years] | 53 [18 to 77] | 51.5 [22 to 81] | 51 [18 to 79] | 52 [18 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 37 | 33 | 109
  Male | 7 | 9 | 13 | 29
Region of Enrollment [Number; unit: participants]
  United States | 46 | 46 | 46 | 138
Right Handedness [Count of Participants; unit: Participants] | 39 | 40 | 44 | 123
College Degree [Count of Participants; unit: Participants] | 21 | 12 | 21 | 54

OUTCOME MEASURES:

1. Primary Outcome: Successful Administration of Naloxone
Description: A successful administration will be defined as administration of the simulated naloxone to the mannequin head or simulated flesh pad within 10 minutes and without any critical errors. Critical errors include: Failure to attach the needle to the syringe, failure to place the device tip into a nostril, failure to remove both caps from the device, failure to remove the cap from the naloxone, failure to depress the device and release the naloxone into the nostril, failure to remove cap from the naloxone, failure to draw up > 90% (0.9 ml) of the naloxone, failure to attach atomizer to the device, failure to puncture the simulated flesh pad with the needle, failure to attach the naloxone to the device, failure to push the naloxone into the simulated flesh pad, drug leakage before administration, and administration of the total volume in a single nostril.
Time Frame: 10 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Intramuscular Administration | Intranasal (Atomizer) | Intranasal (Spray)
Number analyzed (Participants) | 46 | 46 | 46
Participants | 32 | 41 | 46

2. Secondary Outcome: Time to Successful Administration of Naloxone
Description: The time required to successfully administer the simulated naloxone will be reported for each group. Only participants who were successful administering naloxone were included in this analysis.
Time Frame: 10 minutes
Measure: Median (Full Range); unit: Seconds
Arm/Group | Intramuscular Administration | Intranasal (Atomizer) | Intranasal (Spray)
Number analyzed (Participants) | 32 | 41 | 46
Seconds | 99.9 [50 to 420] | 110.3 [68.3 to 288.9] | 34.3 [16.3 to 59.7]

ADVERSE EVENTS:
Arm/Group | Intramuscular Administration | Intranasal (Atomizer) | Intranasal (Spray)
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 0/46 | 0/46 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes